CLINICAL TRIAL: NCT01481844
Title: Sequential Therapy Versus Quadruple Therapy as Second Line Treatment After Failure of the Standard Triple Therapy for H Pylori Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Daniela Munteanu,MD ,Principal Investigator, MD, Principal investigator, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sor006811ctil
Record Dates: First submitted 2011-10-30; First posted 2011-11-30 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Optimization of Second Line Treatment Protocol for H Pylori Eradication
Keywords: sequential therapy; second line treatment; H pylori
MeSH Terms: interventions — Lansoprazole; bismuth subsalicylate; Metronidazole; Tetracycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sequential treatment (Experimental): 1.drugs experimental-Sequential -PPI( Lansoprazole 30mg x2/day) + amoxicillin 1gx2/day for 5days, followed by 5 days of PPI(Lansoprazole 30mg x2/day) + ( Clarithromycin500mg x2/day and Tinidazole 500mg x2/day )
  Interventions: Drug: Lansoprazole , Tab Amoxycillin , Tab Clarithromycin ,Tab Tinidazole
- quadruple therapy (Active Comparator): Quadruple drug regimen (i.e.-14 days of PPI (Lansoprazole 30mg x2/day) + Bismuth Subsalicylate 525mg X4/day + Metronidazole 500mg x3/day + Tetracycline 500mg x4/day )-is standard of care as second line treatment in eradication of H pylori
  Interventions: Drug: Lansoprazole, Bismuth Subsalicylate, Metronidazole, Tetracycline

INTERVENTIONS:
Drug: Lansoprazole , Tab Amoxycillin , Tab Clarithromycin ,Tab Tinidazole — use of Sequential therapy as second line treatment for eradication H pylori currently Sequential therapy is indicated as first line treatment for H pylori eradication
  Arms: sequential treatment
Drug: Lansoprazole, Bismuth Subsalicylate, Metronidazole, Tetracycline — this combination is standard of care as H pylori second line treatment
  Arms: quadruple therapy

SUMMARY:
The aim of this study is to evaluate the efficacy of sequential therapy, i.e. 5 days of PPI + amoxicillin followed by 5 days of PPI + two antimicrobial drugs( clarithromycin and tinidazole ) versus quadruple drug regimen( i.e.-14 days of PPI+ bismuth + metronidazole + tetracycline ) as second line treatment of H. pylori .

DETAILED DESCRIPTION:
a total of 101 patients were randomized to 2 groups : 50 in sequential group and 51 patients in quadruple group . mean age was 43 in both groups. In sequential therapy group 42 patients(84%) completed the treatment , 39 patients returned to follow up . In quadruple group only 33 patients (64.7%) completed the treatment , 29 of them returned to follow up.

Compliance to the treatment was significant better in sequential group comparative to quadruple .Sides effects connected to gastro-intestinal tract were reported in 27(65.9%) of quadruple group patients and in 19(43.2%)of sequential group.

The H pylori was eradicated in 23 of 39 patients in sequential group(59%), and in 19 of the 29 patients in quadruple group(65.5%). no comorbidities like smoking, diabetes or other influenced the efficacy of eradication.

Sequential therapy showed the same eradication rate as second line treatment of H pylori as quadruple one, but was associated with better compliance and less adverse effects.

Both treatments protocols failed to show an appropriate eradication rate in population of Southern Israel .

ELIGIBILITY:
Inclusion Criteria:

1. signed informed consent
2. age at least 18 years
3. persisting H.pylori infection after at least one course of first-line standard triple therapy (Amoxycillin, Clarithromycin or Metronidazole based)

Exclusion Criteria:

1. history of gastrectomy
2. gastric malignancy, including adenocarcinoma and lymphoma
3. previous allergic reaction to antibiotics (amoxicillin, clarithromycin, metronidazole, tetracycline) and proton pump inhibitors
4. Active upper gastrointestinal bleeding within the previous 1 week
5. contraindications to the treatment drugs
6. Pregnant or lactating women
7. Severe concurrent disease or malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The eradication rate after second line treatment based on sequential therapy comparative to eradication rate after second line therapy based on quadriple regimen | 18 month
  H pylori eradication is defined as a negative C-urea breath test 4-16 weeks after completion of tratment.]. (C-urea breath test- Patients are fasted for 4 h before testing. No test meal will be given, and a pre-dose breath sample is obtained. 75 mg of 13C-urea powder dissolved in 50 mL of water is then administered orally, and a second breath sample is collected 30 minutes later. Collected samples are analyzed using an isotope ratio mass spectrometer).

SECONDARY OUTCOMES:
The secondary end points: Adverse effects of sequential and quadruple treatment | 18 months
  -Adverse effects -taste alteration , peripheral neuropathy, seizures, nausea, vomiting, diarrhea, abdominal pain, allergic reaction, photo sensibility-checked at clinical visit by direct question.
compliance with treatment | 18 months
  compliance is considered to be satisfactory when drug intake exceeded 80 %( by pills count).

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Munteanu, MD, Principal Investigator — Soroka UMC
Locations (1):
- Soroca UMC, Beersheba, Israel

REFERENCES:
- [Derived] Munteanu D, Etzion O, Ben-Yakov G, Halperin D, Eidelman L, Schwartz D, Novack V, Abufreha N, Krugliak P, Rozenthal A, Gaspar N, Moshkalo A, Dizingof V, Fich A. Efficacy and safety of sequential versus quadruple therapy as second-line treatment for helicobacter pylori infection-A randomized controlled trial. PLoS One. 2017 Sep 28;12(9):e0183302. doi: 10.1371/journal.pone.0183302. eCollection 2017. PMID 28957341